CLINICAL TRIAL: NCT04004156
Title: Safety Study for An Artificial Disc Replacement "PerQdisc Nucleus Replacement Device" NUCLEUS 181
Brief Title: Safety Study for An Artificial Disc Nucleus Replacement to Treat Chronic Low Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was terminated prematurely due to receipt of CE mark
Sponsor: Spinal Stabilization Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N181
Record Dates: First submitted 2019-06-26; First posted 2019-07-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Degenerative Disc Disease; Chronic Low-back Pain
Keywords: Degenerative Disc Disease; DDD; Chronic Low-back Pain; Low Back Pain; Nucleus Replacement Device; Nucleus Pulposus; Disc Replacement; Back pain; Leg pain; Lumbar Spinal Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain; Back Pain

STUDY DESIGN:
Intervention Model Description: This is an open label study. Patients that are unable to receive an implant due to intraoperative exclusion will receive standard of care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nucleus Replacement (Experimental): All patients that meet the inclusion/exclusion criteria will receive the PerQdisc® Nucleus Replacement Device.
  Interventions: Device: PerQdisc® Nucleus Replacement Device.

INTERVENTIONS:
Device: PerQdisc® Nucleus Replacement Device. — All patients that meet the inclusion/exclusion criteria will receive the PerQdisc® Nucleus Replacement Device.

SUMMARY:
This study will be a prospective, open-label, multi-center study that will collect safety data for the minimally invasive PerQdisc Nucleus Replacement Device deployed to reduce chronic low back pain.

DETAILED DESCRIPTION:
This study will be a prospective, open-label, multi-center study that will collect safety data for the minimally invasive PerQdisc Nucleus Replacement Device (NRD). The NRD is used for surgical replacement of a single nucleus pulposus between spinal lumbar discs L1-S1 using an anterior or lateral transpsoas approach. Currently the surgical gold standard involves spinal fusion of the affected vertebral bodies, reducing range of motion and increasing stress on other vertebral bodies. The goal of nucleus replacement is to reduce chronic low back pain by maintaining disc height while preserving range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Patient is skeletally mature and between 22 and 60 years of age.
* Patient has degenerative disc disease (DDD) at a single level between L1 and S1 as confirmed by:History and clinical findings suggestive of symptomatic DDD, Darkened disc on MRI in T2 weighted images, and decreased disc height (decreased greater than 2 mm compared to adjacent cranial or caudal disc height) with minimum disc height of 6 mm.
* Patient has pre-operative back pain VAS score of greater than or equal to 4 (0-10 scale).
* Patient has pre-operative Oswestry Low Back Disability score of greater than or equal to 40 (0-100 scale).
* Patient has received conservative (non-surgical) treatment for back pain for a minimum of 6 months.
* Patient has signed the approved Informed Consent Form.

Exclusion Criteria:

* Patient has had prior lumbar spine surgery.
* Patient has motion of less than 3 degrees on pre-operative lateral flexion/extension radiographs.
* Patient has ankylosing spondylitis or other spondyloarthropathy.
* Patient has isthmic spondylolisthesis or degenerative spondylolisthesis greater than 2 mm.
* Patient has congenital stenosis or epidural lipomatosis.
* Patient has significant facet disease.
* Patient has any known active malignancy.
* Patient has previously undergone immunosuppressive therapy.
* Patient has active local or system infection.
* Patient has been diagnosed with hepatitis, rheumatoid arthritis, lupus erythematosus, or other autoimmune disease, including AIDS, ARC and HIV
* Patient has diabetes mellitus (Type 1 or 2), requiring daily insulin management.
* Patient has osteopenia of the spine (T-score less than 1.0). All females 45 years of age or older and all males 50 or older should have a DEXA scan to confirm this exclusion.
* Patient has morbid obesity defined as body mass index (BMI) more than 40 or a weight of more than 45 kg (100 lbs) over ideal body weight.
* Patient is pregnant or plans to become pregnant during the course of the study.
* Patient has a known allergy to silicone (polymer and balloon material) or barium sulfate (polymer).
* Patient participated in another investigational drug or device study within the past 30 days.
* Patient belongs to a vulnerable population or has a condition such that his/her ability to provide informed consent, comply with follow-up requirements, or provide self assessments is compromised (e.g. developmentally disables, prisoner, chronic alcohol/ substance abuser)
* Patient has a disc herniation
* Patient has a Schmorl's node in the level to be treated

Intraoperative exclusion criteria:

* Protrusion of the 20A imaging balloon up to or beyond the outer margin of the vertebra during the imaging steps.
* Patient has a violated endplate.
* Patient has a disc space that is too narrow.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Rate of revision surgery at the treated level | 90 days
  Number of patients requiring surgeries to revise the implanted level in the spine divided by the total number of implant surgeries. Express in percentage (0-100)
Rate of expulsion | 90 Days
  The rate of device expulsion. The number of patients determined to have expulsed devices divided by the total number of patients receiving implants.Expressed in percentage (0-100)
Rate of new herniation at the treated level as determined by MRI | 90 days
  Herniation will be determine by MRI. A herniation will be defined as violation of the intervertebral annulus, including expulsion of nucleus material. The response will be yes/no as assessed by the radiologist. Rate will be determined by total number of herniations divided by the total number of implanted devices. Expressed in percentage (0-100)
Rate of new radiculopathy | 90 days
  New complaint of leg pain will be recorded as a yes/no response. Any complaint of new radiculopathy not seen preoperatively. Expressed as total number of new radiculopathy complaints divided by total number of patients. Expressed in percentage (0-100)
MRI assessment of the endplate Modic changes. | 90 days
  Changes to vertebral endplates will be assigned based on Modic classification of I,II or III comparing preoperative grade to grade at 90 days. Possible scores are I,II or III
Rate of surgical procedure technical success | 90 days
  The number of devices successfully implanted divided by the number of successfully devices implanted + unsuccessful implants. Output will be in percentage (0-100)
Improvement in degree of disability as measured by the Oswestry Disability Index (ODI) | 90 days
  Change in absolute Oswestry Index score at 90 days compared to the preoperative score, range is 0-100
Improvement in back pain as measured by 10-centimeter Visual Analog Scale (VAS) | 90 days
  Change in the Visual Analogue Scale (VAS) for back and leg pain on a scale of 0-10 cm comparing preoperative scores to 90 days post-operative.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hess, MD, Study Chair — London Spine Clinic/ATOS-Klinik
Locations (4):
- Onze Lieve Vrouw Ziekenhuis, Aalst, Belgium
- Montreal General Hospital, Montreal, Quebec, Canada
- Clinical Hospital Dubrava, Zagreb, Croatia
- Donauisar Klinikum Deggendorf, Deggendorf, Germany

IPD SHARING:
Plan to Share IPD: No